CLINICAL TRIAL: NCT06399796
Title: Insulin Resistance in Relation to Hyperthyroidism and Hypothyroidism
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Ibrahim Sadek Mohamed, Doctor, Assiut University
Other Study IDs: Thyroid and insulin resistance
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Insulin resistance and its relation to hyperthyrodism and Hypothyroidism

DETAILED DESCRIPTION:
Thyroid hormones (TH) play an important role in regulating energy balance, metabolism of glucose, and lipids. While TH oppose the action of insulin and stimulate the hepatic gluconeogenesis and glycogenolysis they up-regulate the expression of genes such as glucose transporter type-4 (GLUT--4) and phosphoglycerate kinase, involved in glucose transport and glycolysis, respectively, thus acting synergistically with insulin facilitating glucose disposal and utilization in peripheral tissues.

This indicates a possible interplay between thyroid status and insulin sensitivity. Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations. The homeostasis model assessment (HOMA) for IR (HOMA-IR) derives estimates of insulin sensitivity from the mathematical modeling of fasting plasma glucose and insulin concentrations.

Homeostatic model assessment for insulin resistance (HOMA - IR) based on fasting glucose and insulin measurements; derived from the product of the insulin and glucose values divided by a constant, that is, calculated by using the following formula: fasting glucose (mg/dL) X fasting insulin (mU/L) / 405 (for SI units: fasting glucose (mmol/L) X fasting insulin (mU/L) / 22.5) , a value greater than 2 indicates insulin resistance .

In both hyper- as well as hypothyroid groups, there was significant increase in LDL levels. The amount of insulin specifically bound and the number of insulin receptors per cell were inversely correlated with the LDL level. The number of insulin receptors and the amount of insulin bound in the tested subjects with increased LDL were correspondingly low.

ELIGIBILITY:
Inclusion Criteria:

* Adult pations above 18 years old

Exclusion Criteria:

* Any patients with Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on determining the main outcome variable, the estimated minimum required sample size is 108cases (36cases in each group ).
  The sample size was calculated using G*power software 3.1.9.7., based on the following assumptions:
  HbA1C was elevated in 22.3% of hypothyroid group and 21% of hyperthyroid group compared to controls group eleveted only in ( 16.1%) Medium effect size was estimate to be 0.3 Main statistical test is chi_squer test ,goodness of fit Alpha = 0.05, Power = 0.80 Allocation ratio= 1.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of diabetes mellitus among patients with thyroid disorders | baseline
  to prove the prevalence of diabetes mellitus is elevated among patients with thyroid disorders

REFERENCES:
- [Background] Chubb SA, Davis WA, Davis TM. Interactions among thyroid function, insulin sensitivity, and serum lipid concentrations: the Fremantle diabetes study. J Clin Endocrinol Metab. 2005 Sep;90(9):5317-20. doi: 10.1210/jc.2005-0298. Epub 2005 Jun 28. PMID 15985488
- [Background] Raboudi N, Arem R, Jones RH, Chap Z, Pena J, Chou J, Field JB. Fasting and postabsorptive hepatic glucose and insulin metabolism in hyperthyroidism. Am J Physiol. 1989 Jan;256(1 Pt 1):E159-66. doi: 10.1152/ajpendo.1989.256.1.E159. PMID 2643338
- [Background] Clement K, Viguerie N, Diehn M, Alizadeh A, Barbe P, Thalamas C, Storey JD, Brown PO, Barsh GS, Langin D. In vivo regulation of human skeletal muscle gene expression by thyroid hormone. Genome Res. 2002 Feb;12(2):281-91. doi: 10.1101/gr.207702. PMID 11827947
- [Background] Singh BM, Goswami B, Mallika V. Association between insulin resistance and hypothyroidism in females attending a tertiary care hospital. Indian J Clin Biochem. 2010 Apr;25(2):141-5. doi: 10.1007/s12291-010-0026-x. Epub 2010 May 27. PMID 23105900
- [Background] Mari A, Ahren B, Pacini G. Assessment of insulin secretion in relation to insulin resistance. Curr Opin Clin Nutr Metab Care. 2005 Sep;8(5):529-33. doi: 10.1097/01.mco.0000171130.23441.59. PMID 16079624
- [Background] Sanghvi A, Virji MA, Warty V, Dimasi MJ. Differential suppression of lymphocyte cholesterol synthesis by low density lipoprotein and erythrocyte insulin receptors in normolipidemic subjects. Atherosclerosis. 1983 Dec;49(3):307-18. doi: 10.1016/0021-9150(83)90141-7. PMID 6362680